CLINICAL TRIAL: NCT06647212
Title: The Effect of Harmonica Exercises on Cardiorespiratory Exercise Capacity Parameters, Quality of Life and Symptoms of Depression in Patients Undergoing Cardiac Rehabilitation.
Brief Title: Harmonica Exercises for Patients Undergoing Cardiac Rehabilitation.
Acronym: HARMONYCR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katarzyna Piotrowicz (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Piotrowicz, Head of Cardiac Rehabilitation Department, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resolution No.12/24
Record Dates: First submitted 2024-09-29; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; Heart Failure
Keywords: cardiac rehabilitation; harmonica exercises; exercise capacity; quality of life; depression
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Depression

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study arm (Experimental): patients randomized to the study arm will receive a breathing exercise program with standard diatonic mouth harmonica
  Interventions: Other: introducing breathing exercises with the harmonica
- control arm (No Intervention): patients randomized to the control arm will follow standard cardiac rehabilitation program with breathing exercises only

INTERVENTIONS:
Other: introducing breathing exercises with the harmonica — In addition to regular breathing exercises, participants will perform harmonica exercises
  Arms: study arm

SUMMARY:
The study aims to assess the effects of exercises using the harmonica on the exercise capacity, the level of depressive symptoms and disease related quality of life in patients suffering from heart disease attending cardiac rehabilitation program.

The main questions it aims to answer are:

Does harmonica exercise improve exercise capacity in patints with herat disease? Does harmonica exercise affect depression levels and health-related quality of life in patients with heart disease?

Researchers will explore the effect of harmonica exercise on exercise capacity and selected psychological aspects of patients participating in cardiac rehabilitation program

Participants will:

Complete a cardiac rehabilitation program with assessment of exercise capacity at the beginning and end of the program Perform breathing exercises only or breathing exercises and harmonica exercises Keep a diary of their exercises

DETAILED DESCRIPTION:
The project concerns patients with heart diseases participating in a hybrid cardiac rehabilitation program. The hybrid cardiac rehabilitation program takes place in two periods: an initial hospital stay and a main period at home. The initial period allows for the optimization of pharmacotherapy, performing necessary laboratory tests, performing assessment of exercise capacity , planning and conducting training sessions, education focuses on pro-healty behaviours and psychological counseling. The main period is carried out at home and consists of systematic physical training carried out under the supervision of medical personnel.

As part of the effects of cardiac rehabilitation, it is recommended to perform endurance training appropriate to the patient's clinical condition, elements of resistance training and a set of general exercises: including breathing, relaxation, stretching, balance and agility exercises. Breathing exercises are used to improve breathing efficiency and increase the capacity of the respiratory system. The exercises can be performed in a static form, when the patient inhales and exhales in a specific respiratory path, and in a dynamic form, when breathing exercises are combined with movements of the limbs or torso. The training is performed 3-5 times a week for a minimum of 8 weeks, duration is approximately 20-30 minutes. Exercises on the harmonica consist of repeatedly overcoming the very small respiratory resistance created by the instrument during inhalation and exhalation, which results in the generated sound. Therefore - unlike most other wind instruments, which have an adverse effect on the respiratory system - the harmonica was used in exercises for patients with significant respiratory diseases. In the available literature, there are no studies on the use of the harmonica in patients with heart diseases.

One of the most serious and widespread problems of patients with cardiovascular diseases is reduced quality of life and symptoms of depression. Therapy or rehabilitation using music can improve the mental state, sense of self-efficacy and sense of bond with other people, especially among people with symptoms of mood disorders, PTSD or substance abuse. There are no studies on the effect of musical interventions (e.g. using a harmonica) on the somatic and emotional state of people after cardiovascular incidents.

The harmonica exercises were developed by a professional musician, music educator and health sociologist. Duration of a single exercise session: 30 +/- 10 minutes. During the hospital stage, patients will have three lessons with musicians and will receive materials for home exercises. Online communication with musicians will also be possible, in case of doubts about the exercises. Harmonicas used in the study: standard diatonic harmonicas. Principle of exercises: chord playing based primarily on playing rhythms, not melodies, which is the equivalent of exercises for people starting to learn to play the diatonic harmonica.

Patients will receive diaries describing the recommended breathing exercises for the control group and additionally exercises with the harmonica for the study group. In both groups, patients record the amount and time of exercises. After the completion of the rehabilitation cycle, 4-5 weeks, an assessment of the patient's exercise capacity and psychological state will be performed, oriented to refer to the project's goal.

Study type: prospective, randomized, open clinical trial (with a control group) involving patients admitted to a rehabilitation program who express informed consent to participate in the study. Selection to the study or control group will be randomized, after the participant expresses consent to participate.

Study group: patients randomized to the study group were given a breathing exercise program using a standard diatonic mouth harmonica as the only additional element added to the rehabilitation program Control group: patients following standard rehabilitation program Methods: baseline clinical and laboratory data will be collected. To assess physical exercise capacity fallowing will be performed: cardiopulmonary exercise stress test, 6-minute walk test. To assess psychological status the self-reported questionnaires: EQ-5D/ VAS, Brief IPQ-R and PHQ-9 will be administered.

Data collection: The measurements will be taken at randomization and follow-up (the end of rehabilitation cycle).

ELIGIBILITY:
Inclusion Criteria:

patients participating in cardiac rehabilitation program

Exclusion Criteria:

* Decompensated heart failure, with symptoms in NYHA class II-IV within 3 weeks before admission to the Cardiac Rehabilitation Department

  * Poorly controlled hypertension (BP in office measurement >160/100 mmHg)
  * Severe symptomatic heart disease (including valvular);
  * Other severe comorbidities, including those significantly limiting physical performance: chronic kidney disease with GFR <30 ml/min/1.73m2 (according to the CKD-EPI formula), severe form of bronchial asthma/chronic obstructive pulmonary disease (stage C/D ), hypertrophic cardiomyopathy, significant cardiac arrhythmias (persistent/permanent atrial fibrillation, sustained supraventricular/ventricular tachycardia, multiple supraventricular/ventricular extrasystole > 10,000/day), pulmonary embolism in the last 3 months, acute coronary syndrome in the last 7 days, peripheral arterial disease with claudication distance <200 m, generalized active neoplastic process;
  * mental illness/dementia syndrome that prevents full cooperation with the examined person;
  * diseases of the musculoskeletal system that make it impossible to perform an exercise test;
  * contraindications to performing an exercise test;
  * contact allergy to the materials from which the body/cover of the harmonica is made, revealed during exercises
  * lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
exercise capacity | from enrollment to the end of cardiac rehabilitataion at 5 weeks
  Exercise capacity assessed by cardiopulmonary exercise testing measured by peak oxygen consumption.
health related quality of life | from enrollment to the end of cardiac rehabilitataion program at 5 weeks
  Health related quality of life measured by the EuroQOL five dimensions questionnaire.This is a self-reported description of the subject's current health in 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression
symptoms of depression | from enrollment to the end of cardiac rehabilitataion program at 5 weeks
  Syptoms of depressin measured by Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Piotrowicz, MD, PhD, MS, Study Chair — Military Institute of Medicine; Anna Mierzyńska, PhD, MS, Principal Investigator — Military Institute of Medicine
Locations (1):
- Cardiac Rehabilitation Department, Military Institute of Medicine National research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No